CLINICAL TRIAL: NCT01029106
Title: Prospective, Non-Randomized, Observational, Multicentre, Study of the TVT Secur in the Surgical Management of Women With Stress Urinary Incontinence
Brief Title: Gynecare TVT Secur for the Management of Stress Urinary Incontinence (SUI)
Status: Terminated | Type: Observational
Why Stopped: Study design required a change in device
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sender Herschorn, MD, Sunnybrook Health Sciences Centre
Other Study IDs: TVTSecur; 047-2009
Record Dates: First submitted 2009-10-19; First posted 2009-12-09 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Stress Urinary Incontinence
Keywords: SUI; Stress Urinary Incontinence; Patients with Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Gynecare TVT Secur — Implant of the Gynecare TVT Secur

SUMMARY:
This is a prospective, non-randomized, observational, multicentre (5 sites) study in which subjects that have surgically-correctable Stress Urinary Incontinence undergo a TVT SECUR operative procedure.

The study will collect preoperative urologic testing, medical history, and subject quality of life patient questionnaires, Intraoperative procedural data will be collected.

Postoperative complications, urologic, testing, and subject questionnaires will be collected at intervals up to 24 months. The anatomic position of the device will be characterize by transvaginal ultrasound testing.

To determine the rate and/or improvement rate of patients who have received the Gynecare Secur device after 12 months and after 24 months.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible to participate in this study, subjects must meet the following requirements:

1. Subject has agreed to undergo surgical implantation of the TVT SECUR System
2. Subject has the complaint of SUI for at least 6 months prior to the Preoperative Evaluation Visit.
3. Subject has confirmed SUI resulting from urethral hypermobility on cough stress testing.
4. Subject has at least 4 gm of urine leakage on 1-hour pad testing during the Preoperative Screening Visit.
5. Subject is at least 18 years of age to maximum of 85 years of age
6. Subject is willing and able to give written informed consent prior to any study related procedures.
7. Subject is willing to return for follow-up evaluation and questionnaire completion at 4-6 weeks, and at 3, 6, 12 and 24 month follow-ups.
8. Subject is willing to undergo transvaginal ultrasound evaluation at the 4 weeks and 12 month follow-up visit.

Exclusion Criteria:

Subjects will not be eligible for entry into the study if they meet one of the following criteria:

1. Subject is pregnant.
2. Subject has had any previous synthetic sub-urethral sling procedure.
3. Subject has current urinary tract or vaginal infections.
4. Subject has blood coagulation disorders.
5. Subject has a compromised immune system or any other conditions that would compromise healing.
6. Subject has upper urinary tract obstruction.
7. Subject is unwilling to provide written informed consent.
8. Subject is unwilling or unable to return for evaluation at 4-6 weeks, and at 3, 6, 12, and 24 months.
9. Subject has uncontrolled detrusor overactivity.
10. Subject has PVR greater than 100 cc.
11. Subject has Peak Flow Rate less than 10 ml/sec.
12. Subject has urethral diverticulum.
13. Subject has significant pelvic organ prolapse (Grade III/IV) requiring surgical treatment.
14. Subject has had radiation therapy to the pelvic area at any time.
15. Subject has current or active history of pelvic cancer.
16. Subject who in the opinion of the investigator is unable and/or unlikely to comprehend the nature, scope and possible consequences of the study and to follow the study procedures and instructions and complete all study related measurements.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 125 women with SUI from 5 centres across Canada will participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
The primary endpoints are the cure/improvement rate in the cohort at 12 months. | 12 months

SECONDARY OUTCOMES:
Distribution of percentage of subjects having a decrease of pad weight as compared to baseline | 24 months
Decrease in number of pads used within a 24-hour period as compared to baseline | 24 months
Change in patient questionnaires from baseline | 24 months
Change in the sling position on transvaginal ultrasound | 24 months
Cure/improvement rate at 24 months | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sender Herschorn, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada